CLINICAL TRIAL: NCT06301750
Title: A Randomly Controlled Study to Explore Oral vs Nasal Enteral Nutrition Feeding in Alzheimer's Patients
Brief Title: Oral Enteral Nutrition Feeding in Alzheimer's Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad (Other)
Responsible Party: Sponsor-Investigator, Muhammad, Research Director, Ahmadu Bello University Teaching Hospital
Organization: Ahmadu Bello University Teaching Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tube-Alzheimer
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Enteral Nutrition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Oral-esophageal Tube Feeding group (Experimental): This group is hospitalized, while conventional care and enteral nutrition support are provided to the two groups. The Intermittent Oral-esophageal Tube Feeding group receives Intermittent Oral-esophageal Tube Feeding for enteral nutrition support
  Interventions: Behavioral: Conventional Care; Device: Intermittent Oral-esophageal Tube Feeding
- Nasogastric tube group (Active Comparator): This group is hospitalized, while conventional care and enteral nutrition support are provided to the two groups. The Nasogastric tube group receives Nasogastric Tube Feeding for enteral nutrition support
  Interventions: Behavioral: Conventional Care; Device: Nasogastric tube

INTERVENTIONS:
Behavioral: Conventional Care — Basic treatment, including corresponding control of risk factors and education on healthy lifestyles.
  Swallowing training, including lemon ice stimulation, mendelson maneuver, empty swallowing training, and pronunciation training.
  Pulmonary function training, including standing training, cough training, and diaphragm muscle training.
Device: Intermittent Oral-esophageal Tube Feeding — Before each feeding, inside and outside of the tube was cleaned with water. During feeding, the patient should maintain a semi-reclining or sitting position with mouth opened, and the tube was inserted slowly and smoothly into the upper part of the esophagus by medical staffs while the appropriate depth of intubation was checked with the calibration markings on the tube wall. The distance from the incisors to the head part of the tube should be between 22-25 cm. However, the specific depth should be evaluated based on patients' feedback and adjusted accordingly. After insertion, the tail part of the tube should be put into a container full of water and the absence of continuous bubbles indicated a successful intubation. Then, the feeding was to be conducted three times per day with 50 ml per minute and 400-600ml for each feeding.
  Arms: Intermittent Oral-esophageal Tube Feeding group
Device: Nasogastric tube — Within 4 hours after admission, the placement of the feeding tube was conducted by professional medical staffs and after intubation, the tube was secured to the patient's cheek with medical tape. The feeding was conducted once every 3-4 hours, with 200-300ml each time. The total feeding volume was determined based on daily requirements. The feeding content was formulated by the nutritionists based on the patient's condition and relevant guidelines to reach the energy demand as 20-25 kcal/kg/day and protein supplementation of 1.2-2.0 g/kg/day for both two groups. For patients with limited tube feeding compliance, we made appropriate adjustments to ensure that they were not at risk of severe malnutrition as much as possible.
  Arms: Nasogastric tube group

SUMMARY:
This is a prospective multicenter study with Alzheimer's patients with dysphagia. Patients enrolled are randomly divided equally into the observation group and the control group. All patients receive conventional care, and the observation group received Intermittent Oral-esophageal Tube Feeding while the control group received Nasogastric Tube Feeding for enteral nutrition support. Baseline information (demographics, medical history, etc.), nutritional status at admission and after treatment, depression, dysphagia, and quality of life after treatment are compared.

DETAILED DESCRIPTION:
The Alzheimer's disease in the elderly exhibits the high prevalence.This is a prospective multicenter study with Alzheimer's patients with dysphagia. Patients enrolled are randomly divided equally into the observation group and the control group. All patients receive conventional care, and the observation group received Intermittent Oral-esophageal Tube Feeding while the control group received Nasogastric Tube Feeding for enteral nutrition support. Baseline information (demographics, medical history, etc.), nutritional status at admission and after treatment, depression, dysphagia, and quality of life after treatment are compared.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 years and 85 years, meeting the diagnosis of Alzheimer's Disease.
* presence of no contraindication for enteral nutrition.
* with dysphagia verified by Imaging materials.
* with stable vital signs and no severe liver or kidney dysfunction, metabolic disorders, cardiovascular diseases, or multiple complications
* Minimum Mental State Examination ranging from 10-26

Exclusion Criteria:

* unable to cooperate in completing treatment and assessment due to personal reasons or other disorders.
* complicated with other intracranial lesions, such as stroke.
* abnormal structure of swallowing-related organ and tissue.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Level of Hemoglobin | day 1 and day 15
  Hemoglobin was recorded through the blood routine test. (g/L)
Level of Serum albumin | day 1 and day 15
  Serum albumin was recorded through the blood routine test. (g/L)
Level of Total serum protein | day 1 and day 15
  Total serum protein was recorded through the blood routine test. ( g/L)
Level of Serum prealbumin | day 1 and day 15
  Serum prealbumin was recorded through the blood routine test.(g/L)

SECONDARY OUTCOMES:
Body Mass Index | day 1 and day 15
  Body Mass Index was assessed with the combination of body weight and height: weight (kg)/ [height (m)] ^2
Pulmonary Infections | day 1 and day 15
  During the treatment, the occurrence of complications was recorded for both groups. These complications included but were not limited to: 1) Pulmonary Infections: Monitoring for the development of respiratory infections such as pneumonia or bronchitis.
Mini Nutritional Assessment | day 1 and day 15
  Mini Nutritional Assessment is used for assessment of nutritional status, ranging 0 to 30. A higher score indicates the better nutritional status

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Study Chair — Site Coordinator of United Medical Group

IPD SHARING:
Plan to Share IPD: No